CLINICAL TRIAL: NCT00420784
Title: A Phase 2 Study of Telaprevir (VX-950) in Combination With Peginterferon Alfa-2a (Pegasys®), and Ribavirin (Copegus®) in Subjects With Genotype 1 Hepatitis C Who Have Not Achieved Sustained Viral Response With a Prior Course of Interferon Based Therapy
Brief Title: A Study of Telaprevir (VX-950), Pegasys and Copegus in Hepatitis C (PROVE3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX06-950-106
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-07

CONDITIONS: Hepatitis C
Keywords: Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week (Experimental): Single loading dose of telaprevir 1125 milligram (mg) tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily for 12 weeks in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (RBV) tablet orally twice daily at a dose of 1000 milligram per day (mg/day) for subjects weighing less than (<) 75 kilogram (kg) and 1200 mg/day for subjects weighing greater than or equal to (>=) 75 kg, for 24 weeks.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a
- Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week (Experimental): Single loading dose of telaprevir 1125 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily for 24 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 48 weeks.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a
- Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week (Experimental): Single loading dose of telaprevir 1125 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection, for 24 weeks.
  Interventions: Drug: Telaprevir; Drug: Pegylated Interferon Alfa 2a
- PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week (Placebo Comparator): Placebo (PBO) matched to telaprevir tablet orally thrice daily for 24 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 48 weeks.
  Interventions: Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a; Drug: Matching Placebo

INTERVENTIONS:
Drug: Telaprevir — tablet
  Other Names: VX-950
  Arms: Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week; Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week; Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week
Drug: Ribavirin — tablet
  Other Names: RBV
  Arms: PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week; Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week; Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week
Drug: Pegylated Interferon Alfa 2a — Solution for injection
  Other Names: Peg-IFN-alfa-2a
Drug: Matching Placebo — Tablet
  Arms: PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week

SUMMARY:
The PROVE3 trial is a partially double blinded, randomized, Phase 2 research study of an investigational drug, Telaprevir (VX-950) or Placebo, with Pegylated Interferon Alfa 2a (Peg-IFN-alfa-2a, Pegasys®), and Ribavirin (RBV, Copegus®) in people with genotype 1 hepatitis C who have not achieved a Sustained Viral Response (SVR) with a previous treatment of interferon therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 70 years old
* Detectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) greater than or equal to (>=) 10,000 international units per milliliter (IU/mL)
* Must have chronic hepatitis C (genotype 1) and have already received at least one prior course of pegylated interferon alfa 2a with ribavirin
* Cannot also be infected with Human Immunodeficiency Virus or hepatitis B
* Must be judged to be in general good health and able to receive Pegasys® and Copegus®
* No drug or alcohol abuse in the last year
* Must agree to use two effective methods of birth control during the study and for 6 months after you stop taking study medication. One of the methods needs to be a 'barrier' method (condom or diaphragm)
* If you are a woman, you cannot be in this study if you are pregnant or nursing

Exclusion Criteria:

* Participation in any clinical trial of a HCV protease inhibitor of any duration
* Prior response to therapy and failure to achieve SVR which was due to treatment non-compliance
* Any other cause of significant liver disease in addition to hepatitis C; this may include but is not limited to, hepatitis B, drug or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, nonalcoholic steatohepatitis, or primary biliary cirrhosis
* Diagnosed or suspected hepatocellular carcinoma
* History of or current evidence of decompensated liver disease
* Participation in any clinical trial of an investigational drug within 90 days before drug administration or participation in more than 2 drug studies in the last 12 months (exclusive of the current study)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (53):
- United States (41):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - USC, Los Angeles, California
  - Kaiser Permanente Hepatology Research, San Diego, California
  - University of California, San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Englewood, Colorado
  - Bardenton, Florida
  - University of Florida, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Miami, Florida
  - University Hepatitis Center at Bach & Godofsky, Sarasota, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - Virology Treatment Center, Maine Medical Center, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Louis University, St Louis, Missouri
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - New York, New York
  - Durham, North Carolina
  - University Internal Medicine Associates, Inc., Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia Gastroenterology Associates, PA, Columbia, South Carolina
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Liver Institute at Methodist Dallas, Dallas, Texas
  - Advanced Liver Therapies, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Annandale, Virginia
  - Metropolitan Research, Fairfax, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Canada (6):
  - University of Calgary Medical Clinic - Health Science Centre, Calgary, Alberta
  - Edmonton, Alberta
  - BC Hepatitis Program, Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Toronto Western Hospital, Toronto, Ontario
  - Toronto, Ontario
- Germany (2):
  - Universitatsmedizin Berlin, Berlin
  - University Clinic Frankfurt, Department of Internal Medicine, Frankfurt
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus MC University Medical Center, Rotterdam
- Santurce, Puerto Rico

REFERENCES:
- [Derived] Li S, Zhu J, Zhang W, Chen Y, Zhang K, Popescu LM, Ma X, Lau WB, Rong R, Yu X, Wang B, Li Y, Xiao C, Zhang M, Wang S, Yu L, Chen AF, Yang X, Cai J. Signature microRNA expression profile of essential hypertension and its novel link to human cytomegalovirus infection. Circulation. 2011 Jul 12;124(2):175-84. doi: 10.1161/CIRCULATIONAHA.110.012237. Epub 2011 Jun 20. PMID 21690488
- [Derived] McHutchison JG, Manns MP, Muir AJ, Terrault NA, Jacobson IM, Afdhal NH, Heathcote EJ, Zeuzem S, Reesink HW, Garg J, Bsharat M, George S, Kauffman RS, Adda N, Di Bisceglie AM; PROVE3 Study Team. Telaprevir for previously treated chronic HCV infection. N Engl J Med. 2010 Apr 8;362(14):1292-303. doi: 10.1056/NEJMoa0908014. PMID 20375406

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 465 subjects were enrolled, of which 12 subjects discontinued the study prior to study drug administration. A total of 453 subjects started treatment.
Period: Overall Study
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week
Started | 115 | 113 | 111 | 114
Completed | 86 | 55 | 58 | 36
Not Completed | 29 | 58 | 53 | 78
Not completed — Adverse Event | 11 | 29 | 10 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Virologic Stopping Rule | 17 | 26 | 41 | 67
Not completed — Other | 1 | 2 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set = subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week | Total
Number analyzed (Participants) | 115 | 113 | 111 | 114 | 453
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 114 | 111 | 108 | 113 | 446
  >=65 years | 1 | 2 | 3 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (7.8) | 52.0 (5.5) | 51.9 (7.1) | 49.8 (7.2) | 50.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 39 | 38 | 147
  Male | 78 | 80 | 72 | 76 | 306
Region of Enrollment [Number; unit: participants]
  North America | 101 | 103 | 101 | 101 | 406
  Europe | 14 | 10 | 10 | 13 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Undetectable Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Week 24 After the Completion of Study Drug Dosing
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: 24 weeks after the completion of study drug dosing (up to Week 72)
Population: Full Analysis Set = subjects who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week
Number analyzed (Participants) | 115 | 113 | 111 | 114
percentage of participants | 51.3 | 53.1 | 24.3 | 14.0
Statistical Analysis 1: Comparison: Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week vs PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.23, 95% CI 2-sided [4.14 to 16.36]
Statistical Analysis 2: Comparison: Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week vs PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 9.52, 95% CI 2-sided [4.72 to 19.20]
Statistical Analysis 3: Comparison: Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week vs PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week; Test type: Superiority or Other; p = 0.024, Regression, Logistic; Odds Ratio (OR) = 2.31, 95% CI 2-sided [1.12 to 4.75]

2. Secondary Outcome: Percentage of Subjects With Undetectable Plasma HCV RNA at Completion of Study Drug Dosing
Description: as for outcome 1
Time Frame: Completion of study drug dosing (up to Week 48)
Population: Full Analysis Set = subjects who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week
Number analyzed (Participants) | 115 | 113 | 111 | 114
percentage of participants | 75.7 | 67.3 | 54.1 | 29.8

3. Secondary Outcome: Percentage of Subjects With Undetectable Plasma HCV RNA
Description: Percentage of subjects with undetectable HCV RNA at 24 weeks after last dose of study drug for treatment group "PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week" and at 48 weeks after last dose of study drug for treatment groups "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week", "Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week" and "Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week" were presented. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: Up to Week 96 (24 weeks after last dose of study drug for PBO group; 48 weeks after last dose of study drug for telaprevir groups)
Population: Full Analysis Set = subjects who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week
Number analyzed (Participants) | 115 | 113 | 111 | 114
percentage of participants | 48.7 | 44.2 | 22.5 | 14.0
Statistical Analysis 1: Comparison: Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week vs PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.64, 95% CI 2-sided [3.41 to 12.96]
Statistical Analysis 2: Comparison: Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week vs PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.72, 95% CI 2-sided [2.91 to 11.27]
Statistical Analysis 3: Comparison: Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week vs PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week; Test type: Superiority or Other; p = 0.067, Regression, Logistic; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.95 to 4.00]

4. Secondary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any adverse change from the subject's baseline (pre-treatment) condition, including any adverse experience, abnormal recording or clinical laboratory assessment value which occurs during the course of the study, whether it is considered related to the study drug or not. An adverse event includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug. SAE: medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. "Study drug" includes all investigational agents (including placebo, if applicable) administered during the course of the study.
Time Frame: Baseline up to 2 weeks after last dose of study drug (up to Week 50)
Population: Full Analysis Set = subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week
Number analyzed (Participants) | 115 | 113 | 111 | 114
participants
  AEs | 112 | 113 | 105 | 111
  SAEs | 6 | 16 | 6 | 9

5. Secondary Outcome: Number of Subjects With Viral Relapse
Description: Viral relapse was defined as having detectable HCV RNA during antiviral follow-up. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: After last dose of study drug up to 24 week antiviral follow-up (up to Week 72)
Population: Analysis population included subjects who completed their assigned study drug treatment and had undetectable HCV RNA at the completion of treatment (up to Week 48).
Measure: Number; unit: participants
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week
Number analyzed (Participants) | 87 | 76 | 60 | 34
participants | 26 | 10 | 32 | 18

6. Secondary Outcome: Maximum (Cmax), Minimum (Cmin) and Average (Cavg) Plasma Concentration of Telaprevir
Description: Only subjects who received telaprevir were to be analyzed for this outcome. Maximum, minimum and average plasma concentrations observed during assessment period were reported.
Time Frame: Week 2, 4, 8, 12, 16, 24
Population: Pharmacokinetic population included all subjects who provided pharmacokinetic assessments and had evaluable and interpretable data.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Telaprevir: All subjects who received single loading dose of telaprevir 1125 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily for 12 weeks in "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week" reporting group and for 24 weeks in "Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week" and "Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week" reporting groups.
Arm/Group | Telaprevir
Number analyzed (Participants) | 339
nanogram per milliliter (ng/mL)
  Cmax | 2755 (811)
  Cmin | 2335 (733)
  Cavg | 2610 (780)

ADVERSE EVENTS:
Time Frame: Baseline up to 2 weeks after last dose of study drug (up to Week 50)
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week
Serious Adverse Events (participants affected / at risk) | 6/115 | 16/113 | 6/111 | 9/114
Other Adverse Events (participants affected / at risk) | 112/115 | 112/113 | 105/111 | 111/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week (N=115) | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week (N=113) | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week (N=111) | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week (N=114)
Gastroenteritis (Infections and infestations) | 0 | 6 | 3 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Infected insect bite (Infections and infestations) | 0 | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis syndrome (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 6 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 0 | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal tubular acidosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
B-cell unclassifiable lymphoma low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 24 Week (N=115) | Telaprevir 24 Week+Peg-IFN-alfa-2a,RBV 48 Week (N=113) | Telaprevir 24 Week+Peg-IFN-alfa-2a 24 Week (N=111) | PBO 24 Week+Peg-IFN-alfa-2a, RBV 48 Week (N=114)
Fatigue (General disorders) | 77 | 69 | 51 | 64
Influenza like illness (General disorders) | 29 | 36 | 28 | 36
Irritability (General disorders) | 20 | 27 | 16 | 25
Pyrexia (General disorders) | 16 | 27 | 16 | 14
Chills (General disorders) | 17 | 23 | 17 | 15
Injection site erythema (General disorders) | 14 | 10 | 9 | 5
Pain (General disorders) | 8 | 4 | 6 | 4
Oedema peripheral (General disorders) | 3 | 6 | 5 | 1
Nausea (Gastrointestinal disorders) | 41 | 54 | 27 | 39
Diarrhoea (Gastrointestinal disorders) | 37 | 49 | 29 | 22
Haemorrhoids (Gastrointestinal disorders) | 15 | 19 | 14 | 3
Vomiting (Gastrointestinal disorders) | 15 | 13 | 9 | 13
Dry mouth (Gastrointestinal disorders) | 8 | 13 | 9 | 6
Abdominal pain (Gastrointestinal disorders) | 6 | 6 | 7 | 8
Constipation (Gastrointestinal disorders) | 4 | 6 | 2 | 9
Anorectal discomfort (Gastrointestinal disorders) | 8 | 7 | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 7 | 2 | 6
Flatulence (Gastrointestinal disorders) | 6 | 7 | 2 | 3
Proctalgia (Gastrointestinal disorders) | 6 | 1 | 4 | 0
Stomach discomfort (Gastrointestinal disorders) | 7 | 2 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 39 | 50 | 40 | 17
Rash (Skin and subcutaneous tissue disorders) | 43 | 51 | 32 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 16 | 14 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 8 | 12 | 7
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5 | 10 | 6 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 6 | 4 | 7 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 7 | 4 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 6 | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 6 | 2 | 3 | 0
Headache (Nervous system disorders) | 51 | 39 | 40 | 41
Dizziness (Nervous system disorders) | 10 | 20 | 17 | 18
Dysgeusia (Nervous system disorders) | 5 | 10 | 8 | 8
Disturbance in attention (Nervous system disorders) | 7 | 7 | 8 | 7
Memory impairment (Nervous system disorders) | 2 | 8 | 1 | 2
Insomnia (Psychiatric disorders) | 33 | 30 | 20 | 19
Anxiety (Psychiatric disorders) | 10 | 13 | 4 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 16 | 19 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 22 | 15 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | 5 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 6 | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 2 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 3 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 8 | 4 | 3
Urinary tract infection (Infections and infestations) | 5 | 7 | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 30 | 30 | 9 | 9
Neutropenia (Blood and lymphatic system disorders) | 12 | 11 | 8 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5 | 10 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 8 | 5 | 12
Vision blurred (Eye disorders) | 6 | 10 | 7 | 6
Hypertension (Vascular disorders) | 1 | 6 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 22 | 9 | 20
Depression (Psychiatric disorders) | 13 | 17 | 13 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days